CLINICAL TRIAL: NCT07253532
Title: Impact of Vibrotactile Stimulation Via BalanceBelt and IMU-based Gait Analysis in Individuals With Balance Disorders
Brief Title: Vibrotactile Balance Belt Effect on Improving Gait
Acronym: BalanceBelt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00530950
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Hypofunction; Ataxia - Other; Gait Impairment

STUDY DESIGN:
Intervention Model Description: The investigators will have a group of people affected by vestibular disorders. The people affected by vestibular disorders will then be compared to a group of healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Disorders Group with Vibrotactile Stimulation via Balance Belt (Experimental): Participants with balance disorders will wear a vibrotactile stimulation belt (Balance Belt) designed to provide compensatory cues to improve balance and mobility. Physiologic, kinematic, and behavioral responses will be assessed using methods such as the video head impulse test (vHIT), the Dynamic Visual Acuity Test (DVA), and wearable inertial measurement unit (IMU) sensors to measure gait kinematics.
  Interventions: Device: BalanceBelt
- Healthy Controls Group (Age/Gender-Matched Participants Without Balance Disorders) (No Intervention): Participants in the Healthy Controls Group are age- and gender-matched individuals without balance disorders. These participants will serve as a comparison group and will not receive any interventions. The participant's physiologic, kinematic, and behavioral measures will be assessed using the same testing protocols as the experimental group, including the video head impulse test (vHIT), the Dynamic Visual Acuity Test (DVA), and clinical/kinematic evaluations using inertial measurement unit (IMU) sensors.

INTERVENTIONS:
Device: BalanceBelt — The BalanceBelt is a lightweight, wearable device designed to assist individuals with balance impairments. It provides real-time vibrotactile feedback around the waist, which aligns with the user's posture and movements. By delivering sensory cues, the BalanceBelt aids users in maintaining stability and improving awareness of trunk tilt during daily activities. Its non-invasive design allows for continuous use and can be discreetly worn under clothing. The device aims to enhance safety, confidence, and independence for individuals with balance dysfunction, supporting both rehabilitation and long-term mobility improvements.
  Arms: Balance Disorders Group with Vibrotactile Stimulation via Balance Belt

SUMMARY:
This study will examine the effect of using a vibrotactile feedback implemented into a belt, at improving gait in those with gait disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Waist between 60 and 120 cm
* Intact vibration sensitivity around the waist
* Balance disorder and/or a diagnosis of ataxia or vestibular dysfunction (diagnosis based on imaging, clinical and family history, vestibular function tests, and/or genetic testing)
* Speak English

Exclusion Criteria:

* Previous Vestibular Rehabilitation Therapy (VRT) finished less than 2 months ago
* Inability to stand or walk slowly without support in the light on a firm underground
* Neurological, ophthalmological and/or orthopedic disorders that hampers vestibular, oculomotor or gait and posture examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  The Dizziness Handicap Inventory (DHI) is a validated patient-reported outcome measure designed to assess the perceived impact of dizziness on daily function. It includes 25 items categorized into physical, emotional, and functional domains, with responses scored on a scale from 0 (no impact) to 100 (maximum impact). Higher scores indicate greater disability.
Activities Balance Confidence Scale (ABC) | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  The Activities Balance Confidence Scale (ABC) is a validated self-reported questionnaire designed to measure an individual's confidence in maintaining balance during various daily activities, such as walking on uneven surfaces, climbing stairs, or reaching overhead. The scale consists of 16 items, with each activity rated on a percentage scale from 0% (no confidence) to 100% (complete confidence). Higher scores indicate greater balance confidence.
Bilateral Vestibular Questionnaire (BVQ) | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  The Bilateral Vestibular Questionnaire (BVQ) is a 54-item patient-reported outcome measure designed to assess the range of symptoms experienced by individuals with bilateral vestibular dysfunction and the impact on daily life. The questionnaire evaluates seven domains: imbalance, oscillopsia, other physical symptoms, cognition, emotion, behavioral changes and limitations, and social life. Each item is scored on a six-point Likert scale ranging from "never" to "always." Score range 0-324. Higher scores reflect greater symptom severity and reduced quality of life.
Single-Item and Visual Analog Scales (VAS) | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  Single-item measures and Visual Analog Scales (VAS) will be used to assess specific aspects of participants' experiences and treatment responses. Each scale involves a numerical or visual rating system typically ranging from 0 to 10, or 0 to 100, depending on the domain being assessed. These scales measure variables such as limitations in daily life, perceived health, expectations for future recovery, and the overall effectiveness of previous rehabilitation therapies. A higher score indicates more positive outcomes or perceptions.
Video Head Impulse Test (vHIT) | Baseline, 3 weeks, 1-2-3-4 months
  The Video Head Impulse Test (vHIT) is a clinical test used to assess the vestibulo-ocular reflex (VOR) by measuring eye movement responses to head rotations. This test evaluates the function of the three semicircular canals, providing insight into vestibular physiology. During the test, participants wear video goggles that record eye movements while the head is gently rotated to either side at a velocity of ~150°/s, consistent with standardized vHIT protocols. The primary outcome measure is VOR gain (eye velocity/head velocity), with lower gain values potentially indicating vestibular dysfunction.
Dynamic Visual Acuity (DVA) | Baseline, 3 weeks, 1-2-3-4 months
  The Dynamic Visual Acuity (DVA) test is a validated clinical measure used to assess the ability to maintain clear vision during head movements. The test evaluates the vestibulo-ocular reflex (VOR) by comparing static visual acuity (head stationary) with visual acuity during dynamic head rotations in the horizontal and vertical planes (e.g., head movements right, left, up, and down). Participants are seated 2 meters from the testing screen, and head rotation speeds must reach a minimum of 80°/s to generate the randomized optotype. The primary measure is logMAR (logarithm of the minimum angle of resolution) scores, where higher logMAR values indicate worse visual acuity during movement.
Functional Gait Assessment (FGA) | Baseline, 3 weeks, 1-2-3-4 months
  The Functional Gait Assessment (FGA) is a clinical tool used to evaluate gait performance in individuals during different walking tasks. It consists of 10 tasks, including walking while changing speeds, walking with head turns, walking backward, stepping over obstacles, and walking in tandem. Each task is scored on a 0-3 scale, with a total score range of 0-30 indicating optimal performance, and lower scores reflecting greater balance impairments and reduced gait functionality. The FGA is validated for identifying fall risk. Scores below 22/30 indicate fall risk in older adults.
Timed Up and Go (TUG) | Baseline, 3 weeks, 1-2-3-4 months
  The Timed Up and Go (TUG) test is a validated tool for assessing functional mobility and fall risk. Participants are instructed to rise from a seated position, walk 3 meters, turn 180°, walk back, and return to a seated position. The time taken to complete the sequence is recorded as the primary outcome. Faster times indicate normal functional mobility, while slower times (>13.5 seconds for older adults) are indicative of increased fall risk, particularly in individuals with vestibular disorders.
Timed Up and Go Dual Task | Baseline, 3 weeks, 1-2-3-4 months
  The Timed Up and Go Dual Task test is a dual-task modified version of the traditional TUG protocol, which further assesses the impact of cognitive load on mobility and balance. Participants perform the same tasks as the TUG test (stand, walk 3 meters, turn, and return to sit) while simultaneously counting backwards from 100 by threes (or another similar cognitive challenge). Timings exceeding 15 seconds in elderly individuals are associated with increased fall risk.
Gait Velocity (10-Meter Walk Test) | Baseline, 3 weeks, 1-2-3-4 months
  Gait velocity will be measured using the 10-Meter Walk Test (10MWT), a validated assessment tool for evaluating walking speed during a self-selected comfortable pace over a short distance. Participants will be instructed to walk 10 meters while gait speed is recorded, with or without an assistive device as appropriate. The average speed (meters/second) is calculated and will be used as the primary outcome measure.
Sway energy and sway over time (Adaptation Test) | Baseline, 3 weeks, 1-2-3-4 months
  The Adaptation Test assesses participants' ability to maintain stability and adapt to unexpected changes in surface tilt. Testing is conducted using a rotating force plate, which provides controlled motion stimuli in two directions: toes-up and toes-down. Participants will stand on the force plate while wearing the Virtualis Motion (VR) headset, which provides immersive visual environments to simulate balance challenges and enhance sensorimotor engagement. Postural stability is evaluated by measuring sway energy, which quantifies force and the extent of anterior-posterior sway, as well as sway over time, which measures center of pressure (COP) movement across the duration of the trials. These measures provide insight into a participant's balance control and adaptive strategies during repeated tilt trials.

SECONDARY OUTCOMES:
Oscillopsia Functional Index (OFI) | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  The Oscillopsia Functional Index (OFI) is a 43-item patient-reported outcome measure designed to quantify the functional impact of oscillopsia symptoms on various activities of daily living. Participants rate level of difficulty across tasks such as walking, riding in a car, recognizing faces, and navigating environments. Each item is scored on a scale from 0 (no symptoms or difficulty) to 5 (unable to perform the activity due to symptoms), with additional options for marking activities as "not applicable." Total OFI scores range from 0 to 215, with higher scores indicating greater impairment.
Falls Efficacy Scale - International (FES-I) | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  The Falls Efficacy Scale - International (FES-I) is a widely validated self-reported questionnaire designed to assess a participant's concern about falling during a variety of daily physical and social activities. It consists of 16 items covering tasks performed both inside and outside the home, such as cleaning, shopping, and walking. Each item is rated on a 4-point Likert scale ranging from "Not at all concerned" (1) to "Very concerned" (4), resulting in a total score range of 16-64, with higher scores indicating greater concerns about falling.
EQ-5D-5L Quality of Life Questionnaire | Baseline, 3 weeks, 1-2-3-4-5-11-23-35 months
  The EQ-5D-5L is a standardized instrument for measuring health-related quality of life. It evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on five levels ranging from "no problems" to "extreme problems," creating a profile of a participant's health status. Additionally, participants complete a Visual Analog Scale (VAS) to rate overall health from 0 ("worst imaginable health") to 100 ("best imaginable health").
Vestibular Evoked Myogenic Potential (VEMP) | Baseline, 3 weeks, 1-2-3-4 months
  The Vestibular Evoked Myogenic Potential (VEMP) test is a clinical measure used to assess the function of the vestibular system, focusing specifically on the otolith organs (utricle and saccule). VEMP includes two types: cervical VEMP (cVEMP), which assesses saccular function through responses from the sternocleidomastoid neck muscle, and ocular VEMP (oVEMP), which evaluates utricular function through responses from the orbicularis oculi eye muscles. Participants are positioned reclined and equipped with electrodes over the relevant muscles. Auditory stimuli, such as clicks or tone bursts, are delivered via earphones to each ear individually, and participants are asked to lift the head (cVEMP) or look upward (oVEMP) to optimize muscle activation. Test results include latency and amplitude of evoked potential responses, with reduced or absent responses indicating possible vestibular dysfunction.
Vestibular Nystagmogram (VNG) | Baseline, 3 weeks, 1-2-3-4 months
  The Vestibular Nystagmogram (VNG) is a standard clinical test used to evaluate the function of the vestibular system, particularly the horizontal semicircular canal. It involves recording participants' eye movements while wearing video goggles designed to track nystagmus (involuntary eye movements) in response to various stimuli. Participants follow an infrared light with the eyes during certain conditions, and nystagmus responses are evaluated after exposure to both cold air and warm air stimuli administered into the ear canal.
Scale for Ocular Motor Disorders in Ataxia (SODA) | Baseline, 3 weeks, 1-2-3-4 months
  The Scale for Ocular Motor Disorders in Ataxia (SODA) is a clinical rating tool designed to quantify and characterize ocular motor dysfunction in patients with cerebellar ataxia and related disorders. SODA systematically evaluates a range of oculomotor deficits, including gaze-holding and smooth pursuit abnormalities, saccadic dysmetria (hypometria and hypermetria), saccade velocity and restriction, gaze-evoked and spontaneous nystagmus (horizontal and vertical), saccadic oscillations, and abnormalities in the vestibulo-ocular reflex (VOR). Each domain is scored based on the observed severity and type of deficit. Higher SODA scores correspond to more severe ocular motor dysfunction.
Dynamic Gait Index (DGI) | Baseline, 3 weeks, 1-2-3-4 months
  The Dynamic Gait Index (DGI) is a validated clinical tool used to assess gait, balance, and fall risk during dynamic walking tasks. The DGI includes 8 tasks, such as walking while changing speeds, turning the head, stepping over obstacles, and pivoting. Each task is scored on a 0-3 scale, with a total maximum score of 24 indicating optimal performance, and lower scores reflecting greater gait and balance impairments. A score below 19/24 indicates a significantly increased risk of falls (2.58 times greater likelihood of falling within the previous 6 months).
Scale for the Assessment and Rating of Ataxia (SARA) | Baseline, 3 weeks, 1-2-3-4 months
  The Scale for the Assessment and Rating of Ataxia (SARA) is a validated clinical tool designed to quantify the severity of ataxia symptoms. SARA consists of 8 tasks that evaluate various aspects of motor function, including gait, stance, sitting, and limb coordination (such as finger chase, nose-finger tests, and heel-shin tests). Each task is rated on a 0-4 scale, with total scores ranging from 0 (no ataxia) to 40 (most severe ataxia). Lower scores reflect minimal impairment, while higher scores indicate greater dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Millar, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kingma H, Hougaard DD, van de Berg R. Subconscious vibrotactile stimulation improves mobility and balance in patients with bilateral vestibulopathy: adherence over 2 years. Front Neurol. 2024 Oct 8;15:1491195. doi: 10.3389/fneur.2024.1491195. eCollection 2024. PMID 39440249
- [Background] Kingma H, Felipe L, Gerards MC, Gerits P, Guinand N, Perez-Fornos A, Demkin V, van de Berg R. Vibrotactile feedback improves balance and mobility in patients with severe bilateral vestibular loss. J Neurol. 2019 Sep;266(Suppl 1):19-26. doi: 10.1007/s00415-018-9133-z. Epub 2018 Dec 5. PMID 30519776
- [Background] Hegeman J, Honegger F, Kupper M, Allum JH. The balance control of bilateral peripheral vestibular loss subjects and its improvement with auditory prosthetic feedback. J Vestib Res. 2005;15(2):109-17. PMID 15951624
- [Background] Dozza M, Chiari L, Horak FB. Audio-biofeedback improves balance in patients with bilateral vestibular loss. Arch Phys Med Rehabil. 2005 Jul;86(7):1401-3. doi: 10.1016/j.apmr.2004.12.036. PMID 16003671
- [Background] Chiari L, Dozza M, Cappello A, Horak FB, Macellari V, Giansanti D. Audio-biofeedback for balance improvement: an accelerometry-based system. IEEE Trans Biomed Eng. 2005 Dec;52(12):2108-11. doi: 10.1109/TBME.2005.857673. PMID 16366234
- [Background] Guyot JP, Perez Fornos A, Guinand N, van de Berg R, Stokroos R, Kingma H. Vestibular assistance systems: promises and challenges. J Neurol. 2016 Apr;263 Suppl 1:S30-5. doi: 10.1007/s00415-015-7922-1. Epub 2016 Apr 15. PMID 27083882
- [Background] Beylergil SB, Karmali F, Wang W, Bermudez Rey MC, Merfeld DM. Vestibular roll tilt thresholds partially mediate age-related effects on balance. Prog Brain Res. 2019;248:249-267. doi: 10.1016/bs.pbr.2019.04.019. Epub 2019 May 24. PMID 31239136
- [Background] Lucieer F, Vonk P, Guinand N, Stokroos R, Kingma H, van de Berg R. Bilateral Vestibular Hypofunction: Insights in Etiologies, Clinical Subtypes, and Diagnostics. Front Neurol. 2016 Mar 4;7:26. doi: 10.3389/fneur.2016.00026. eCollection 2016. PMID 26973594
- [Background] Starkov D, Strupp M, Pleshkov M, Kingma H, van de Berg R. Diagnosing vestibular hypofunction: an update. J Neurol. 2021 Jan;268(1):377-385. doi: 10.1007/s00415-020-10139-4. Epub 2020 Aug 7. PMID 32767115
- [Background] van Stiphout L, Szmulewicz DJ, Guinand N, Fornos AP, Van Rompaey V, van de Berg R. Bilateral vestibulopathy: a clinical update and proposed diagnostic algorithm. Front Neurol. 2023 Dec 19;14:1308485. doi: 10.3389/fneur.2023.1308485. eCollection 2023. PMID 38178884
- See also: Website of the BalanceBelt device — https://balancebelt.net/en/